CLINICAL TRIAL: NCT00927641
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of HKT-500 in the Treatment of Pain Associated With Mild to Moderate Ankle Sprain
Brief Title: HKT-500 in the Treatment of Adult Patients With Ankle Sprain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hisamitsu Pharmaceutical Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HKT-500-US17
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Ankle Sprain
Keywords: Ankle Sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketoprofen Patch (HKT-500) (Active Comparator): Two Ketoprofen HKT-500 patches applied to target ankle once daily for 14 days
  Interventions: Drug: Ketoprofen Patch
- Placebo Patch (Placebo Comparator): Two placebo patches placed on target ankle once daily for 14 days
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: Ketoprofen Patch — Two Ketoprofen HKT-500 patches applied to target ankle once daily for 14 days
  Other Names: Topical Patch
  Arms: Ketoprofen Patch (HKT-500)
Other: Placebo Patch — Two placebo patches placed on target ankle once daily for 14 days
  Other Names: Sham treatment
  Arms: Placebo Patch

SUMMARY:
The objective of this study is to demonstrate the multiple-dose efficacy and safety of HKT-500 for the treatment of ankle sprain.

DETAILED DESCRIPTION:
A Randomized, Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of HKT-500 in the Treatment of Pain Associated With Mild to Moderate Ankle Sprain

ELIGIBILITY:
Inclusion Criteria:

* mild to Moderate Ankle Sprain

Exclusion Criteria:

* Any women of childbearing potential who has a positive urine pregnancy test, who is lactating, who is not surgically sterile (by tubal ligation or hysterectomy), who is not at least 2 years postmenopausal, or has not practiced an acceptable form of birth control (defined as the use of an intrauterine device with spermicide, a barrier method with spermicide, condoms with spermicide, subdermal implant, oral contraceptives, or abstinence) for at least 2 months prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change from the baseline of the 100-mm VAS pain intensity score during monopodal weight bearing for 1 second at Visit 3 (Day 3 + 1 day) | 3 days + 1

SECONDARY OUTCOMES:
Assessment of the subject's VAS pain intensity during monopodal weight bearing, at rest and in motion, summed pain intensity difference at rest and in motion, cumulative effect of pain reduction | 14 days

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Hisamitsu Investigator Site, Birmingham, Alabama
  - Hisamitsu Investigator Site, Phoenix, Arizona
  - Hisamitsu Investigator Site, Tucson, Arizona
  - Hisamitsu Investigator Site, Hot Springs, Arkansas
  - Hisamitsu Investigator Site, Anaheim, California
  - Hisamitsu Investigator Site, Buena Park, California
  - Hisamitsu Investigator Site, Long Beach, California
  - Hisamitsu Investigator Site, San Diego, California
  - Hisamitsu Investigator Site, San Luis Obispo, California
  - Hisamitsu Investigator Site, Daytona Beach, Florida
  - Hisamitsu Investigator Site, Hialeah, Florida
  - Hisamitsu Investigator Site, Jacksonville, Florida
  - Hisamitsu Investigator Site, Lauderdale Lakes, Florida
  - Hisamitsu Investigator Site, Oldsmar, Florida
  - Hisamitsu Investigator Site, Ormond Beach, Florida
  - Hisamitsu Investigator Site, South Miami, Florida
  - Hisamitsu Investigator Site, Evansville, Indiana
  - Hisamitsu Investigator Site, Omaha, Nebraska
  - Hisamitsu Investigator Site, Blackwood, New Jersey
  - Hisamitsu Investigator Site, South Bound Brook, New Jersey
  - Hisamitsu Investigator Site, Johnson City, Tennessee
  - Hisamitsu Investigator Site, Dallas, Texas
  - Hisamitsu Investigator Site, West Valley City, Utah
  - Hisamitsu Investigator Site, Danville, Virginia